CLINICAL TRIAL: NCT04682093
Title: Risk Stratification of Patients With Suspected COVID-19 Presenting to the ED (EUROCOV Study)
Brief Title: Risk Stratification of Patients With Suspected COVID-19 Presenting to the ED
Acronym: EUROCOV
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: European Society for Emergency Medicine (EUSEM) Research Network (Network)
Responsible Party: Sponsor
Other Study IDs: 123456
Record Dates: First submitted 2020-12-22; First posted 2020-12-23 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Covid19
Keywords: Covid19; Emergencies; epidemiology; prognosis
MeSH Terms: conditions — COVID-19; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project is an unfunded collaboration of approximately 30 emergency departments across Europe led by the EUSEM research network. It involves collection of data in relation to determining the epidemiology and outcome of adult patients who present to emergency departments with a suspected Covid infection.

DETAILED DESCRIPTION:
Over the past 6 months, the world has faced a novel infection disease outbreak, due to a novel coronavirus, the severe acute respiratory syndrome coronavirus (SARS-CoV2), with a massive impact on healthcare resource.

In Europe, numbers of confirmed cases continue to rise. Europe is currently one of the regions with the highest number of Covid-19 cases and deaths due to this emergent diseases.

Most COVID-19 infected patients present with mild to moderate acute respiratory symptoms, including cough, fever, dyspnea and pneumonia. About 20% will present with severe or critical manifestations of the disease, including pneumonia, respiratory failure and acute respiratory distress syndrome (ARDS).

Anticipating the needs for hospitalization in ward and/or intensive care is crucial.

Emergency departments are at the front line for triaging patients with suspected Covid-19 and referring them to the appropriate level of care.

In Europe, the number of ED patients with suspected Covid-19 is variable; rate of hospitalization from ED reaches 40% for this population.

Risk stratification and management decisions of patients presenting to the ED with suspected COVID-19 is a challenge for emergency physicians.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>= 18 years old) attending the ED with a clinical suspicion of COVID-19 based on the presence of the following criteria
* Fever >= 38 °C
* respiratory symptoms (dyspnea, cough, expectorations)
* any other symptoms suggestive of COVID-19 including digestive signs (diarrhea, anosmia…)

Exclusion Criteria:

* None

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Adult patients (>= 18 years old) attending the ED with a clinical suspicion of COVID-19 based on the presence of the following criteria
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
hospitalization | 30 days
  hospitalization after ED visit
length of hospital stay | 30 days
  Hospital LOS
in-hospital mortality | 30 days
  Death during hospitalization
ICU admission | 30 days
  ICU admission after ED visit

CONTACTS AND LOCATIONS:
Overall Officials: Said LARIBI, MD, PhD, Principal Investigator — EUSEM Research network chair
Locations (5):
- EUSEM RN Country lead, Zagreb, Croatia
- EUSEM RN Country lead, Hämeenlinna, Finland
- EUSEM RN Country lead, Tours, France
- EUSEM RN Country lead, Athens, Greece
- EUSEM RN Country lead, Forlì, Italy

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Young BE, Ong SWX, Kalimuddin S, Low JG, Tan SY, Loh J, Ng OT, Marimuthu K, Ang LW, Mak TM, Lau SK, Anderson DE, Chan KS, Tan TY, Ng TY, Cui L, Said Z, Kurupatham L, Chen MI, Chan M, Vasoo S, Wang LF, Tan BH, Lin RTP, Lee VJM, Leo YS, Lye DC; Singapore 2019 Novel Coronavirus Outbreak Research Team. Epidemiologic Features and Clinical Course of Patients Infected With SARS-CoV-2 in Singapore. JAMA. 2020 Apr 21;323(15):1488-1494. doi: 10.1001/jama.2020.3204. PMID 32125362